CLINICAL TRIAL: NCT00623116
Title: Kallmann Syndrome in Finland
Brief Title: A Study to Characterize Epidemiology, Clinical and Genetic Features of Kallmann Syndrome in Finland
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital for Children and Adolescents, Finland (Other)
Responsible Party: Taneli Raivio, MD, Ph D, Hospital for Children and Adolescents, Helsinki University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 231408; 286/E7/2007
Record Dates: First submitted 2008-01-11; First posted 2008-02-25 (Estimated); Last update posted 2008-02-25 (Estimated); Status verified 2008-01

CONDITIONS: Kallmann Syndrome
Keywords: Kallmann Syndrome; hypogonadotropic hypogonadism
MeSH Terms: conditions — Kallmann Syndrome; Hypogonadism | interventions — Gonadotropins; Estrogens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Short withdrawal of testosterone, gonadotropins or estrogenic compounds (see below) — clinical examination, biochemical profile, and genetic characterization. Possibility to stop hormone therapy with drugs containing testosterone (Atmos®, Testim®, Testogel®, Nebido®, Panteston®, Sustanon®), FSH (Gonal-F®, Puregon®), hCG (Pregnyl®), estrogenic compounds (such as Estrofem®, Divigel®, Estrena®, Climara®, Estradot®, Evorel®, Femseven®: Merimono®, Progynova®, Ovestin®, Zumenon®, Estrogel®, Femoston®, Femoston combi®, Divina®, Divitren®, Indivina®, Estalis sekvens®, Evorel sequi®, Novofem®, Trisekvens®, Activelle®, Estalis®, Evorel conti®, Kliogest®, Mericomb®, Mericomb Mite®, Merigest®: Angeliq®) for 3 mo to assess reversibility of GnRH-deficiency will be offered.

SUMMARY:
Objective is to characterize epidemiology, clinical and genetic features of Kallmann syndrome in Finland.

DETAILED DESCRIPTION:
Kallmann syndrome is comprised of idiopathic hypogonadotropic hypogonadism and anosmia (inability to smell). Associated phenotypes may include cryptorchidism, microphallus, bone deformations, mirror movements, hearing loss and infertility. Objective is to characterize epidemiology, clinical and genetic features of Kallmann syndrome in Finland.

ELIGIBILITY:
Inclusion Criteria:

* Kallmann syndrome
* Age 15 yrs or more

Exclusion Criteria:

* Severe mental retardation

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-12; Primary Completion 2012-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Clinical features including quality of life, reversibility and genetic features of Kallmann syndrome in Finland | 0, 3 mo and during subsequent F/U

SECONDARY OUTCOMES:
epidemiology | by 2012 (anticipated)

CONTACTS AND LOCATIONS:
Overall Officials: Taneli J Raivio, MD PhD, Study Director — Hospital for Children and Adolescents, Helsinki University Central Hospital
Locations (1):
- Hospital for Children and Adolescents, Helsinki University Central Hospital, Helsinki, Finland